CLINICAL TRIAL: NCT05694962
Title: Low-Dose Radiation Therapy for Severe COVID-19 Pneumonia: A Multicenter Phase II Prospective Randomized Controlled Study
Brief Title: Low-Dose Radiation Therapy for Severe COVID-19 Pneumonia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Collaborators: Nanjing Chest Hospital (Unknown); The Affiliated BenQ Hospital of Nanjing Medical University (Unknown); Central South University (Other); Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Dr. He Xia, Vice President, Jiangsu Cancer Institute & Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LDRT-SCov19
Record Dates: First submitted 2023-01-20; First posted 2023-01-23 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19; Radiation Therapy; Pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): supportive care and standard of care drug therapies (i.e., glucocorticosteroids, Paxlovid, etc.) plus 1.5Gy single treatment of whole-lung radiation therapy
  Interventions: Radiation: Low-Dose Radiation Therapy
- Control group (No Intervention): supportive care and standard of care drug therapies (i.e., glucocorticosteroids, Paxlovid, etc.)

INTERVENTIONS:
Radiation: Low-Dose Radiation Therapy — 1.5Gy single treatment of whole-lung radiation therapy
  Arms: Treatment group

SUMMARY:
This phase II trial studies low-dose radiation therapy as a treatment for patients with severe COVID-19 pneumonia to improve clinical status.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare treatment of severe COVID-19 pneumonia between supportive care and standard of care drug therapies versus supportive care and standard of care drug therapies plus low-dose, whole-lung radiation therapy

OUTLINE:

Patients undergo 1.5Gy of single low-dose radiation therapy. After completion of study treatment, patients are followed up at days 1-7, and 14 after last dose of intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Have had a positive test confirming the diagnosis of COVID-19;
2. Have had clinical signs of severe acute respiratory syndrome or pneumonia (dyspnea, cough, with need for oxygen support at the time of enrollment);
3. Have visible consolidations/ground glass opacities on chest x-ray or computed tomography;
4. Have been on ventilator support for no longer than 5 calendar days prior to the schedule date of delivery of low-dose radiation therapy;
5. They voluntarily participate in this clinical trial, gave informed consent and signed the informed consent form.

Exclusion Criteria:

1. Have received chest radiotherapy before
2. Bacteria, fungi and other infections other than novel coronavirus infection;
3. Combined with severe primary diseases such as cardiovascular, cerebrovascular, liver, kidney, hematopoietic and endocrine system or immune system diseases (the upper limit of liver function ALT and AST> normal reference value, the upper limit of Scr> normal reference value, poor blood glucose control);
4. Mental retardation, mental disorders;
5. Planned pregnancy, pregnancy, lactation women and during the trial;
6. Allergy constitution or allergy to the drug ingredients and excipients of this test;
7. Participated in other clinical trials in the recent 1 month;
8. The Investigator does not considered appropriate to participate in this clinical trial.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement | 28 days after radiation therapy
  improvement of oxygen saturation in percentage

SECONDARY OUTCOMES:
Temperature | 28 days after radiation therapy
  Temperature in degrees (˚C)
Heart Rate | 28 days after radiation therapy
  Heart rate in beats per minutes
Systolic blood pressure | 28 days after radiation therapy
  Systolic blood pressure in mm Hg Systolic blood pressure in mm Hg
Respirations Respirations Respirations Respirations Respirations Respirations | 28 days after radiation therapy
  Respiratory rate in breaths per minute
FiO2 | 28 days after radiation therapy
  Fi02 in percentage
PEEP Tidal volume Tidal volume | 28 days after radiation therapy
  Positive end expiratory pressure (PEEP) in cm H20
Overall survival Overall survival | 28 days after radiation therapy
  Survival in percentage
Chest CT can | 28 days after radiation therapy
  CT scans with volume of consolidation measured in cubic centimeters
Blood Test | 28 days after radiation therapy
Urine Test | 28 days after radiation therapy

IPD SHARING:
Plan to Share IPD: No